CLINICAL TRIAL: NCT05476952
Title: The Effect of Lean Body Weight-adjusted Rocuronium Dose on Intubation Conditions: a Prospective Observational Study
Brief Title: Lean Body Weight-adjusted Rocuronium Dose and Intubation Conditions
Acronym: LBW
Status: Completed | Type: Observational
Sponsor: DUYGU DEMİROZ (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, DUYGU DEMİROZ, Principal Investigator, Inonu University
Organization: Inonu University (Other)
Other Study IDs: Inonu universty OF MEDİCİNE
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Body Weight Changes; Rocuronium; Intubation Conditions
Keywords: the lean body weight, rocuronium, intubation conditions
MeSH Terms: conditions — Body Weight Changes | interventions — bis(p-chlorophenyl)acetic acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with a normal weight between 18.5 and 24.9 BMI Groups will be divided into 2 groups by their own luck. According to DDA, rocuronium will be evaluated as "DDA", and group numbers given according to TBW will be evaluated as "K".
  Interventions: Procedure: he patients who are administered rocuronium according to LBW were categorized as "LBW", and The group number for those administer according to TBW was categorized as "K".
- Group 2: overweight patients with a BMI between 25-29.9 Groups will be divided into 2 groups by their own luck. According to DDA, rocuronium will be evaluated as "DDA", and group numbers given according to TBW will be evaluated as "K".
  Interventions: Procedure: he patients who are administered rocuronium according to LBW were categorized as "LBW", and The group number for those administer according to TBW was categorized as "K".
- Group 3: patients with a BMI of 30-34.9 in obesity class 1 Groups will be divided into 2 groups by their own luck. According to DDA, rocuronium will be evaluated as "DDA", and group numbers given according to TBW will be evaluated as "K".
  Interventions: Procedure: he patients who are administered rocuronium according to LBW were categorized as "LBW", and The group number for those administer according to TBW was categorized as "K".

INTERVENTIONS:
Procedure: he patients who are administered rocuronium according to LBW were categorized as "LBW", and The group number for those administer according to TBW was categorized as "K". — Patients will be divided equally and validly by the one who will be placed in opaque sealed envelopes on a self-paid basis. One group will be given 0.6 mg/kg rocuronium on an LBW basis (Curon ® 50 mg/5 mL [Mustafa Nevzat, Istanbul, Turkey]), and the other group will be given 0.6 mg/kg rocuronium on a TBW basis.
  Other Names: Groups will be divided into 2 groups by their own luck. According to DDA, rocuronium will be evaluated as "DDA", and group numbers given according to TBW will be evaluated as "K".

SUMMARY:
In this study, researchers wiil administer rocuronium, based on either the lean body weight or the total body weight in patients with body mass index (BMI) of 18.5 to 34.9 and compared the duration of action of the drug and its effects on tracheal intubation conditions and hemodynamic parameters..

DETAILED DESCRIPTION:
The whole body will be routinely monitored with electrocardiogram, oximetry oximetry, and non-invasive arterial monitoring. For anesthesia induction, intravenous (IV) fentanyl 50-100 µg and propofol 2mg/kg will be ventilated 100% by lightning. After optimal general anesthesia was achieved, the ulnar nerve was adapted and monitored at the wrist with TOF-Watch® SX (Organon, Swords Co., Dublin, Ireland). LBW lower content of 0.6 mg/kg rocuronium will be administered. K subgrade similar a dose based on TBW will be administered. The time to duration of rocuronium TOF responses will be measured (T1 (seconds)). All consumers will be intubated with a Macintosh laryngoscope diameter with endotracheal sold with inner tubes of 7.5 8.0 mm and 7 mm to 7.5 mm. A single air anesthetist will evaluate the intubation target according to the Han-Raulo intubation scoreboard. Anesthesia will be provided with sevoflurane and an additional dose of phenyl. Monitoring with TOF was continued until the initial fasciculation power (T2=min) of the adductor pollicis decreased to 25% and was approached to an additional rocuronium dose of 0.3mg/kg. All anesthetic agents for operation will be discontinued and extubated when the TOF value reaches 90%.

ELIGIBILITY:
Inclusion Criteria:

Patients who will receive general anesthesia Operations that will take less than 6 hours Patients to be provided with rocuronium neuromuscular blockade

Exclusion Criteria:

Renal, hepatic, neuromuscular, and metabolic diseases Craniotomies, cardiac, thoracic, and large vessel surgeries Those who did not want to participate in the study will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-65 years, with ASA (American Society of Anesthesiologists physical status) ≤ II
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate intubation conditions with LBW adjusted rocuronium dose . | 3 mount
  MAINTAINING SUFFICIENT INTUBATION CONDITIONS WITH LOW DOSE ROCURONIUM

CONTACTS AND LOCATIONS:
Overall Officials: duygu demiröz, Study Director — INONU UNİVERSİTY
Locations (1):
- Inonu universitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasold KL, Parks AC, Phelan DML, Pontifex MB, Pivarnik JM. Reliability and Validity of Commercially Available Low-Cost Bioelectrical Impedance Analysis. Int J Sport Nutr Exerc Metab. 2019 Jul 1;29(4):406-410. doi: 10.1123/ijsnem.2018-0283. PMID 30507268
- [Background] Erstad BL, Barletta JF. Dosing of neuromuscular blocking agents in patients with obesity: A narrative review. Anaesth Intensive Care. 2021 Mar;49(2):98-104. doi: 10.1177/0310057X20968573. Epub 2021 Apr 27. PMID 33906465
- [Derived] Demiroz D, Colak YZ, Iclek SK, Erdogan MA, Yagci NA, Durmus M, Gulhas N. Does Rocuroinum Dose Adjusted Due to Lean Body Weight Provide Adequate Intubation Conditions?: A Prospective Observational Study. Int J Clin Pract. 2022 Oct 5;2022:6840960. doi: 10.1155/2022/6840960. eCollection 2022. PMID 36263238